CLINICAL TRIAL: NCT04626596
Title: A Phase 3, Open-label, Multi-center, Single Arm Study to Assess Contraceptive Efficacy and Safety of the Etonogestrel (MK-8415) Implant During Extended Use From 3 Years After Insertion in Females 35 Years of Age or Younger
Brief Title: A Study to Assess Contraceptive Efficacy and Safety of Etonogestrel (ENG) Implant Beyond 3 Years of Use (MK-8415-060)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 8415-060; 2020-001232-95 (EudraCT Number); MK-8415-060 (Other: Merck)
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-02

CONDITIONS: Contraception
MeSH Terms: interventions — Endoglin; Drug Implants; etonogestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- ENG implant (Experimental): Participants will have the ENG 68 mg implant inserted and in place for 36 months before enrollment. The ENG implant will remain in place for an additional 24 months.
  Interventions: Combination Product: Radiopaque Etonogestrel (ENG) Implant

INTERVENTIONS:
Combination Product: Radiopaque Etonogestrel (ENG) Implant — 68 mg subdermal implant
  Other Names: Org 32222; Nexplanon; Implanon-NXT; SCH900415; MK-8415

SUMMARY:
The primary purpose of this study is to assess the efficacy and safety of the etonogestrel (ENG) contraceptive implant during participants' fourth and fifth years of use when used as the only method of contraception. The ENG implant is currently approved for a 3-year duration, and this study aims to confirm available evidence suggesting that the ENG implant remains highly effective when used up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Not diagnosed with perimenopause or menopause.
* Heterosexually active with a partner who is not known to be subfertile, sterilized, or infertile, and is seeking contraception for pregnancy.
* Palpable intact ENG implant in the upper inner-arm for 36 months from the date of insertion at the time of enrollment, and has documentation of the insertion date (for example, Nexplanon user card or medical record completed on the date of insertion).
* Does not desire a pregnancy within the 24 months after enrollment, is willing to continue use of the implant for an additional 24 months, and is not intending to use any other form of contraception (eg, condoms) from enrollment until after implant removal at 24 months post enrollment.
* Good physical and mental health in the medical judgment of the investigator.
* History of regular menstrual cycles of 21 to 35 days before the insertion of the ENG implant or before hormonal contraceptive use (which may have preceded the current implant use).
* Able and willing to adhere to all required study procedures, including study visits and eDiary entries, and not planning to relocate during the study.

Exclusion Criteria:

* Conceived a pregnancy during use of the current implant or a past contraceptive implant.
* Known or suspected pregnancy at the time of screening or enrollment visit.
* History of subfertility or infertility.
* Breastfeeding.
* Untreated gonorrhea, chlamydia, or trichomonas or symptomatic vaginitis/cervicitis.
* Significantly abnormal cervical cytology (Pap) or pathology results either at screening or documented in the 36-month period prior to enrollment.
* Current use of an intrauterine device/intrauterine system (IUD/IUS).
* Presence of more than one ENG implant.
* Use of daily/monthly hormonal contraceptives, sex steroids, or GnRH agonist/antagonist within 3 months prior to enrollment.
* Use of injectable hormonal contraceptive with 3-month duration within 9 months prior to enrollment.
* Use of injectable GnRH agonist with 3-month duration within 10 months prior to enrollment .
* Use of medications that induce liver enzymes within 2 months prior to enrollment.
* Untreated or unresolved vaginal bleeding or spotting attributable to underlying pathology in the 12 months before screening.
* Frequent, prolonged, or excessive vaginal bleeding/spotting in the 12 months prior to screening which has not been evaluated to detect underlying pathology.
* History of venous thromboembolism or arterial thromboembolism, transient ischemic attack, angina pectoris, or claudication.
* Any condition associated with an increased risk of venous thromboembolism.
* Uncontrolled or severe hypertension at screening visit.
* Clinically significant liver disease, including active viral hepatitis or cirrhosis.
* History of malignancy within 5 years before screening, except treated skin cancer.
* History of sex steroid-influenced malignancies (eg, genital organs, breasts).
* History or presence of liver tumors (benign or malignant).
* Known allergy/sensitivity or contraindication to the ENG implant or lidocaine with epinephrine.
* History of drug or alcohol abuse or dependence within 24 months prior to enrollment. Routine use of alcohol or marijuana that is not considered abuse or dependence is not exclusionary.
* Use of an investigational drug within 2 months prior to enrollment. Long-term follow up of an investigational compound for COVID-19 is allowed 2 months after the last administered dose.
* Staff or immediate family members of the investigational site or Sponsor directly involved with this study.

Max Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 498 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Pregnancy Rate (Pearl Index) for At Risk Cycles During Extended-Duration Use | Up to 24 months
  The Pearl Index is expressed as the number of on-treatment pregnancies per 100 woman-years of exposure. An on-treatment pregnancy is defined as a confirmed pregnancy with an estimated date of conception 36 months to 60 months since the date of implant insertion. Exposure in 100 woman-years is equal to the number of cycles of use/1300, and one woman-year is defined as a period of 13 treatment cycles, each 28 days long. Only "at risk" cycles for conception will be included in this Pearl Index calculation. An at risk cycle is defined as a cycle during which participants with ENG implant had affirmed heterosexual intercourse without the use of additional contraception.
Pregnancy Rate (Pearl Index) for Alternative At Risk Cycles During Extended-Duration Use | Up to 24 months
  The Pearl Index is expressed as the number of on-treatment pregnancies per 100 woman-years of exposure. An on-treatment pregnancy is defined as a confirmed pregnancy conceived with an estimated date of conception 36 months to 60 months since the date of implant insertion. Exposure in 100 woman-years is equal to the number of cycles of use/1300, and one woman-year is defined as a period of 13 treatment cycles, each 28 days long. Only "alternative at risk" cycles will be included in this Pearl Index calculation. An alternative at risk cycle is defined as a cycle in which participants with ENG implant did not use additional contraception, but without the requirement for affirmed heterosexual intercourse.
Number of Participants Who Experience One or More Adverse Events During Extended-Duration Use | Up to approximately 27 months
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Number of Participants Who Discontinue Treatment (Implant Removed) Due to an Adverse Event During Extended-Duration Use | Up to approximately 24 months
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.

SECONDARY OUTCOMES:
Pregnancy Rate (Pearl Index) for At Risk Cycles During Year 4 of Implant Use | Up to 12 months
  Pearl Index will be calculated as the number of on-treatment pregnancies per 100 woman-years of exposure. Exposure in 100 woman-years is equal to the number of cycles of use/1300, and one woman-year is defined as a period of 13 treatment cycles, each 28 days long. Only "at risk" cycles for conception will be included in this Pearl Index calculation. An at risk cycle is defined as a cycle during which participants with ENG implant had affirmed heterosexual intercourse without the use of additional contraception.
Pregnancy Rate (Pearl Index) for At Risk Cycles During Year 5 of Implant Use | Up to 12 months
  Pearl Index will be calculated as the number of on-treatment pregnancies per 100 woman-years of exposure. Exposure in 100 woman-years is equal to the number of cycles of use/1300, and one woman-year is defined as a period of 13 treatment cycles, each 28 days long. Only "at risk" cycles for conception will be included in this Pearl Index calculation. An at risk cycle is defined as a cycle during which participants with ENG implant had affirmed heterosexual intercourse without the use of additional contraception.
Cumulative Pregnancy Rate During 5 Years of Implant Use | Up to 60 months (From 3 years prior to study entry to 2 years after study entry)
  Cumulative on-treatment pregnancy rate will be calculated based on life table analysis over 5 years of implant use.
Cumulative Pregnancy Rate During 4 Years of Implant Use | Up to 48 months (From 3 years prior to study entry to 1 year after study entry)
  Cumulative on-treatment pregnancy rate will be calculated based on life table analysis over 4 years of implant use.
Pregnancy Rate (Pearl Index) for At Risk Cycles During 5 Years of Implant Use | Up to 60 months (From 3 years prior to study entry to 2 years after study entry)
  Pearl Index will be calculated as the number of on-treatment pregnancies per 100 woman-years of exposure. Exposure in 100 woman-years is equal to the number of cycles of use/1300, and one woman-year is defined as a period of 13 treatment cycles, each 28 days long. Only "at risk" cycles for conception will be included in this Pearl Index calculation. An at risk cycle is defined as a cycle during which participants with ENG implant had affirmed heterosexual intercourse without the use of additional contraception. The number of at-risk cycles of use for each of the 3 years prior to study entry will be estimated.
Pregnancy Rate (Pearl Index) for Alternative At Risk Cycles During 5 Years of Implant Use | Up to 60 months (From 3 years prior to study entry to 2 years after study entry)
  Pearl Index will be calculated as the number of on-treatment pregnancies per 100 woman-years of exposure. Exposure in 100 woman-years is equal to the number of cycles of use/1300, and one woman-year is defined as a period of 13 treatment cycles, each 28 days long. Only "alternative at risk" cycles will be included in this Pearl Index calculation. An alternative at risk cycle is defined as a cycle in which participants with ENG implant did not use additional contraception, but without the requirement for affirmed heterosexual intercourse. The number of alternative at risk cycles of use for each of the 3 years prior to study entry will be estimated.
Number of Bleeding Days During Extended-Duration Use as Assessed in 90-day Reference Periods | Up to 24 months
  Participants will record daily vaginal bleeding in an electronic diary. A bleeding day is defined as any day (24 hours) with bloody vaginal discharge requiring more than one sanitary product (i.e., pad, panty liner, tampon, or menstrual cup) or, if only a menstrual cup is used, more than 5 mL of blood accumulates. Number of bleeding days will be assessed per 90-day reference period (RP).
Number of Spotting Days During Extended-Duration Use as Assessed in 90-day Reference Periods | Up to 24 months
  Participants will record daily vaginal spotting in an electronic diary. A spotting day is defined as any day (24 hours) with bloody vaginal discharge requiring at most one sanitary product (i.e. pad, panty liner, tampon, or menstrual cup containing 5 ml [inclusive] or less of blood). Number of spotting days will be assessed per 90-day reference period (RP).
Number of Bleeding and/or Spotting Days During Extended-Duration Use as Assessed in 90-day Reference Periods | Up to 24 months
  Participants will record daily vaginal bleeding and/or spotting in an electronic diary. A bleeding day is defined as any day (24 hours) with bloody vaginal discharge requiring more than one sanitary product (i.e., pad, panty liner, tampon, or menstrual cup) or, if only a menstrual cup is used, more than 5 mL of blood accumulates. A spotting day is defined as any day (24 hours) with bloody vaginal discharge requiring at most one sanitary product (i.e. pad, panty liner, tampon, or menstrual cup containing 5 ml [inclusive] or less of blood). Number of bleeding and/or spotting days will be assessed per 90-day reference period (RP).
Mean Length of Bleeding and/or Spotting Episodes During Extended-Duration Use as Assessed in 90-day Reference Periods | Up to 24 months
  Participants will record daily vaginal bleeding and/or spotting in an electronic diary (eDiary). A bleeding day is defined as any day (24 hours) with bloody vaginal discharge requiring more than one sanitary product (i.e., pad, panty liner, tampon, or menstrual cup) or, if only a menstrual cup is used, more than 5 mL of blood accumulates. A spotting day is defined as any day (24 hours) with bloody vaginal discharge requiring at most one sanitary product (i.e. pad, panty liner, tampon, or menstrual cup containing 5 ml [inclusive] or less of blood). A bleeding and/or spotting episode is defined as one or more consecutive days during which bleeding and/or spotting is recorded in the eDiary, bounded bleeding/spotting-free days.
Percentage of Participants per 90-day Reference Period with Amenorrhea During Extended-Duration Use | Up to 24 months
  Participants will record daily vaginal bleeding and/or spotting in an electronic diary (eDiary). Amenorrhea is defined as no bleeding or spotting recorded in the eDiary per 90-day reference period (RP).
Percentage of Participants per 90-Day Reference Period with Infrequent Bleeding and/or Spotting During Extended-Duration Use | Up to 24 months
  Participants will record daily vaginal bleeding and/or spotting in an electronic diary (eDiary). A bleeding day is defined as any day (24 hours) with bloody vaginal discharge requiring more than one sanitary product (i.e., pad, panty liner, tampon, or menstrual cup) or, if only a menstrual cup is used, more than 5 mL of blood accumulates. A spotting day is defined as any day (24 hours) with bloody vaginal discharge requiring at most one sanitary product (i.e. pad, panty liner, tampon, or menstrual cup containing 5 ml [inclusive] or less of blood). Infrequent bleeding and/or spotting is defined as less than 3 episodes of bleeding and/or spotting per 90-day reference period (RP).
Percentage of Participants per 90-Day Reference Period with Frequent Bleeding and/or Spotting During Extended-Duration Use | Up to 24 months
  Participants will record daily vaginal bleeding and/or spotting in an electronic diary (eDiary). A bleeding day is defined as any day (24 hours) with bloody vaginal discharge requiring more than one sanitary product (i.e., pad, panty liner, tampon, or menstrual cup) or, if only a menstrual cup is used, more than 5 mL of blood accumulates. A spotting day is defined as any day (24 hours) with bloody vaginal discharge requiring at most one sanitary product (i.e. pad, panty liner, tampon, or menstrual cup containing 5 ml [inclusive] or less of blood). Frequent bleeding and/or spotting is defined as more than 5 episodes of bleeding and/or spotting per 90-day reference period (RP).
Percentage of Participants per 90-Day Reference Period with Normal Frequency Bleeding and/or Spotting During Extended-Duration Use | Up to 24 months
  Participants will record daily vaginal bleeding and/or spotting in an electronic diary (eDiary). A bleeding day is defined as any day (24 hours) with bloody vaginal discharge requiring more than one sanitary product (i.e., pad, panty liner, tampon, or menstrual cup) or, if only a menstrual cup is used, more than 5 mL of blood accumulates. A spotting day is defined as any day (24 hours) with bloody vaginal discharge requiring at most one sanitary product (i.e. pad, panty liner, tampon, or menstrual cup containing 5 ml [inclusive] or less of blood). Normal frequency of bleeding and/or spotting is defined as 3 to 5 episodes of bleeding and/or spotting per 90-day reference period (RP).
Percentage of Participants per 90-Day Reference Period with Prolonged Bleeding and/or Spotting During Extended-Duration Use | Up to 24 months
  Participants will record daily vaginal bleeding and/or spotting in an electronic diary (eDiary). A bleeding day is defined as any day (24 hours) with bloody vaginal discharge requiring more than one sanitary product (i.e., pad, panty liner, tampon, or menstrual cup) or, if only a menstrual cup is used, more than 5 mL of blood accumulates. A spotting day is defined as any day (24 hours) with bloody vaginal discharge requiring at most one sanitary product (i.e. pad, panty liner, tampon, or menstrual cup containing 5 ml [inclusive] or less of blood). Prolonged bleeding and/or spotting is defined more than 14 continuous days of bleeding and/or spotting, per 90-day reference period (RP).
Number of Complications Associated with Implant Removal | Up to 24 months
  Complications associated with implant removal will include failed implant removal; implant site fibrosis; extension of incision of >1 cm; removal of a nonpalpable implant; removal of a deeply placed implant; implant removal in an operating room; implant removal requiring general anesthesia; implant removal requiring regional anesthesia; implant removal requiring imaging guidance; nerve injury during implant removal; vascular injury during implant removal; other complications of device removal not previously mentioned.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Lead, Study Director — Organon and Co
Locations (67):
- United States (64):
  - Alabama Clinical Therapeutics (Site 0222), Birmingham, Alabama
  - Desert Star Family Planning (Site 0193), Phoenix, Arizona
  - Precision Trials (Site 0187), Phoenix, Arizona
  - Visions Clinical Research Tucson (Site 0134), Tucson, Arizona
  - Essential Access Health (Site 0163), Los Angeles, California
  - Matrix Clinical Research Inc (Site 0105), Los Angeles, California
  - University of California Los Angeles (Site 0119), Los Angeles, California
  - University of California, Davis (Site 0124), Sacramento, California
  - Stanford University (Site 0112), Stanford, California
  - Planned Parenthood of the Rocky Mountains (Site 0196), Denver, Colorado
  - Comprehensive Womens Health Center (Site 0194), Denver, Colorado
  - Physicians' Research Options, LLC (Site 0166), Lakewood, Colorado
  - University Of Florida (Site 0144), Jacksonville, Florida
  - Emerald Coast Obstetrics and Gynecology (Site 0203), Panama City, Florida
  - Lenus Research & Medical Group Llc (Site 0102), Sweetwater, Florida
  - Comprehensive Clinical Trials LLC (Site 0101), West Palm Beach, Florida
  - Mount Vernon Clinical Research (Site 0111), Sandy Springs, Georgia
  - Rosemark (Site 0177), Idaho Falls, Idaho
  - Planned Parenthood of Illinois (PPIL) (Site 0200), Chicago, Illinois
  - Indiana University (Site 0220), Indianapolis, Indiana
  - McFarland Clinic, PC (Site 0217), Ames, Iowa
  - Cypress Medical Research Center (Site 0226), Wichita, Kansas
  - Southern Clinical Research Associates (Site 0219), Metairie, Louisiana
  - Johns Hopkins Bayview Medical Center (Site 0225), Baltimore, Maryland
  - Boston University Medical Center (Site 0167), Boston, Massachusetts
  - Planned Parenthood League of Massachusetts (Site 0135), Boston, Massachusetts
  - Michigan Medicine (Site 0108), Ann Arbor, Michigan
  - Saginaw Valley Medical Research Group, LLC (Site 0198), Saginaw, Michigan
  - Planned Parenthood of North Central States (PPNCS) (Site 0113), Minneapolis, Minnesota
  - Metro Jackson OBGYN/SKYCRNG (Site 0233), Jackson, Mississippi
  - Planned Parenthood of the Saint Louis Region & Southwest Missouri (Site 0158), St Louis, Missouri
  - Washington University (Site 0129), St Louis, Missouri
  - Office of Edmond Pack, MD (Site 0168), Las Vegas, Nevada
  - Capital Health OB/GYN- Lawrenceville (Site 0190), Lawrenceville, New Jersey
  - Albuquerque Clinical Trials (Site 0210), Albuquerque, New Mexico
  - Bosque Women's Care (Site 0211), Albuquerque, New Mexico
  - Icahn School of Medicine at Mount Sinai (Site 0155), New York, New York
  - Columbia Univ. Medical Center (Site 0118), New York, New York
  - Montefiore Medical Center (Site 0103), The Bronx, New York
  - Carolina Women's Research and Wellness Center (Site 0154), Durham, North Carolina
  - Eastern Carolina Women's Center (Site 0159), New Bern, North Carolina
  - Velocity Clinical Research, Cincinnati (Site 0230), Cincinnati, Ohio
  - The Ohio State University (Site 0176), Columbus, Ohio
  - HWC Women's Research Center (Site 0199), Englewood, Ohio
  - Oregon Health Sciences University Hospital (Site 0128), Portland, Oregon
  - OB/GYN Associates of Erie (Site 0183), Erie, Pennsylvania
  - University of Pittsburgh - Magee Womens Hospital (Site 0100), Pittsburgh, Pennsylvania
  - Palmetto Clinical Research (Site 0133), Summerville, South Carolina
  - University of Tennessee Medical Center Knoxville (Site 0218), Knoxville, Tennessee
  - Gadolin Research (Site 0232), Beaumont, Texas
  - Signature Gyn Services (Site 0201), Fort Worth, Texas
  - Planned Parenthood of the Gulf Coast (Site 0106), Houston, Texas
  - University of Texas Health Science Center (Site 0178), Houston, Texas
  - Centex Studies, Inc. (Site 0171), Houston, Texas
  - Advances in Health, Inc. (Site 0209), Pearland, Texas
  - Tekton Research - Floyd Curl Drive (Site 0228), San Antonio, Texas
  - Physicians' Research Options, LLC (Site 0204), Pleasant Grove, Utah
  - JBR Clinical Research (Site 0174), Salt Lake City, Utah
  - Tidewater Clinical Research Inc (Site 0162), Norfolk, Virginia
  - Eastern Virginia Medical School (Site 0146), Norfolk, Virginia
  - Multicare Health System Institute for Research and Innovation (Site 0188), Cheney, Washington
  - Seattle Women's: Health, Research, Gynecology (Site 0149), Seattle, Washington
  - Planned Parenthood Great Northwest, Hawai'i, Alaska, Indiana, Kentucky (Site 0110), Seattle, Washington
  - North Spokane Women's Clinic (Site 0137), Spokane, Washington
- Puerto Rico (3):
  - Advance Medical Concept PSC (Site 0313), Cidra, PR
  - Clinical Research Puerto Rico Inc (Site 0302), San Juan, PR
  - FDI Clinical Research (Site 0305), San Juan, PR

IPD SHARING:
Plan to Share IPD: No